CLINICAL TRIAL: NCT01028937
Title: Hyperopia Correction Using the NTK Optimal Keratoplasty (Opti-K) System
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: NTK Enterprises, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTK-1
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Results first posted 2019-05-09 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-04

CONDITIONS: Hyperopia
Keywords: Hyperopia correction; Laser vision correction; Optimal keratoplasty
MeSH Terms: conditions — Hyperopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hyperopia (Experimental): The NTK Optimal Keratoplasty System/Procedure is indicated for the temporary improvement of distance uncorrected visual acuity (in patient eyes that have manifest refraction, spherical equivalent equal to +1.0 to +2.5 Diopters, with less than or equal to 0.75 Diopters of refractive astigmatism (minus cylinder format) and with uncorrected distance visual acuity less than 20/40 but greater than or equal to 20/80. Patients must be at least 40 years of age with a documented stability of refraction for the prior 12 months, as demonstrated by a change of less than or equal to 0.5 Diopters in MRSE. The magnitude of D-UCVA improvement by Opti-K treatment may diminish over time, caused by some regression of effect in addition to natural progressive loss of accommodation and, for most patients, progressive hyperopic shift with increasing age.
  Interventions: Device: Optimal Keratoplasty

INTERVENTIONS:
Device: Optimal Keratoplasty — Laser treatment in 16 spots at treatment energy densities up to 48 mJ per spot

SUMMARY:
The purpose of this U.S. Clinical Trial on treatment of sighted eyes is to investigate the safety and effectiveness of optimal keratoplasty (Opti-K™) treatments for hyperopia correction using the NTK Enterprises (NTK) Opti-K System.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment is limited to subjects who satisfy the following inclusion criteria:

  * Male or Female
  * Any race
  * Patient is at least 40 years old.
  * Patient has bilateral sight with at least one eye with low hyperopia [with +1.0 to +2.75 D spherical component of manifest refraction, less than or equal to 0.75 D cylindrical component of manifest refraction (minus cylinder format) and manifest refraction, spherical equivalent of +1.0 to +2.5 D].
  * Patient has documented stable refraction defined as a change in baseline MRSE of ≤ 0.5 D for the 12 month period prior to primary Opti-K Tx as verified by consecutive refractions, medical records or prescription history.
  * Patient is able to tolerate full cycloplegic refraction while not under cycloplegia.
  * Patient has distance uncorrected visual acuity (D-UCVA) less than 20/40 and better than or equal to 20/80 in both eyes.
  * Patient has stable D-UCVA as documented by a change of ≤ 1 line of D-UCVA for the 12 month period prior to baseline measurements.
  * Patient has distance and near best spectacle corrected visual acuity (D-BSCVA and N-BSCVA) of 20/40 or better in both eyes.
  * Patient has normal videokeratography (i.e., without distorted or unclear corneal mires).
  * Contacts lens wearers must:

    1. discontinue use of soft or gas permeable contact lenses at least two weeks prior to baseline measurements or discontinue use of hard or rigid gas permeable contact lenses at least three weeks prior to baseline measurements and
    2. have two central keratometry readings and two manifest refractions taken at least one week apart that do not differ by more than 0.5 D in either meridian; mires should be regular.
  * Patient is willing and able to comply with all pre-treatment and follow-up requirements, including the ability to read English to complete the NEI-RQL questionnaire.
  * Patient understands the nature of the procedure, as well as potential\ risks or limitations of the treatment, and provides informed consent

Exclusion Criteria:

* Patients are not permitted to enroll in the study if they meet any of the following exclusion criteria:

  * Patients with latent hyperopia > 1.0 D (i.e., baseline MRSE and CRSE should not differ by more than 1.0 D)
  * Patients with nystagmus
  * Patients with previous intraocular or corneal surgery
  * Patients with any residual, recurrent or active ocular disease or corneal abnormality, including any of the following: corneal diameter < 9 mm; central corneal thickness < 500 µm; mild to severe dry eye disease; uncontrolled uveitis; severe blepharitis; lagophthalmos; glaucoma; intraocular pressure > 21 mm Hg; cataract; history of uveitis;corneal shape disorders (keratoconus, keratoglobus, pellucid marginal degeneration, significant irregular corneal astigmatism, etc.);history of herpes zoster/simplex keratitis
  * Patients with cloudy cornea or cloudy anterior chamber
  * Patients with allergy to anesthetics or postoperative medications
  * Patients with chronic allergic reactions, tearing and/or ocular irritation
  * Patients who are hypersensitive to pain stimulus
  * Patients taking systemic medications (NSAIDs, etc.) that affect wound healing
  * Patients taking amiodarone, isotretinoin and/or sumatriptan
  * Patients requiring administration of topical or systemic ophthalmic medications other than the study medications - use of corticosteroids or antimetabolites is specifically contraindicated.
  * Patients with a recent history (within one week prior to treatment) of using ophthalmic medications containing preservatives (benzalkonium chloride,etc.) and/or other ocular drugs that are cytotoxic
  * Patients who are immunocompromised (by, for example, infectious diseases such as HIV, herpes, etc. and/or by immunosuppressive medications) or who have autoimmune diseases such as lupus, rheumatoid arthritis, etc.
  * Patients with diabetes
  * Pregnant, planning to be pregnant or lactating women
  * Patients with unusual hormonal status due to, for example, hormone replacement therapy
  * Patients who have taken or who plan to take oral contraceptives within one year prior to, or following, treatment
  * Patients with unrealistic expectations
  * Patients participating in other ophthalmic clinical trials during this clinical investigation
  * Persons who, in the determination of the investigator, are not competent to understand the procedure or the actions asked of them as research subjects
  * Persons who may not be able to complete the requirements of returning to the investigator's clinic over the period of the study, or who may be difficult to locate or contact on short notice. This does not preclude vacations or travel.
  * Persons who cannot achieve corneal applanation using the SAWSR device or cannot tolerate application of the SAWSR device or who cannot remain motionless for at least 5 seconds after verifying proper SAWSR mounting.
  * Patients who are likely to be exposed to high levels of ultraviolet radiation(from sunlight, tanning lights, etc.) without protective eyewear during the one year period following Opti-K treatment

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-12; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Lockerman, Study Director — NTK Enterprises
Locations (1):
- Laser Vision Medical Associates, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hyperopia
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Hyperopia: Hyperopia treatment
Arm/Group | Hyperopia
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.8 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: The Proportion of Eyes (Target: at Least 85%) That Achieve Successful Distance Uncorrected Visual Acuity (D-UCVA) Improvement Defined as 2 Lines (10 Letters) or More Improvement in D-UCVA Following Tx Will be Reported.
Description: The proportion of eyes (target: at least 85%) that achieve successful distance uncorrected visual acuity (D-UCVA) improvement defined as 2 lines (10 letters) or more improvement in D-UCVA following Tx will be reported
Time Frame: 1 year post-treatment
Population: Eyes
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Groups:
- Treatment Group: Eyes that underwent Opti-K treatment
Arm/Group | Treatment Group
Number analyzed (Participants) | 5
Number analyzed (Eyes) | 5
Eyes | 4

2. Secondary Outcome: The Proportion of Eyes That Achieve Distance Uncorrected Visual Acuity (D-UCVA) of 20/40 or Better Following Tx and the Proportion of Eyes That Achieve D-UCVA of 20/40 or Better as a Function of the Pre-Tx D-UCVA Will Both be Reported.
Description: The proportion of eyes that achieve distance uncorrected visual acuity (D-UCVA) of 20/40 or better following Tx and the proportion of eyes that achieve D-UCVA of 20/40 or better as a function of the pre-Tx D-UCVA will both be reported.
Time Frame: 1 year post-treatment
Population: 1 year follow-up
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Treatment Group
Number analyzed (Participants) | 5
Number analyzed (Eyes) | 5
Eyes | 5

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Hyperopia
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-06): https://cdn.clinicaltrials.gov/large-docs/37/NCT01028937/Prot_SAP_000.pdf